CLINICAL TRIAL: NCT00965146
Title: An Open Label, Post-market, Non-randomized, Multi-center Study of the Outcomes of the Scorpio® Cruciate Retaining (CR) Total Knee System
Brief Title: Scorpio® Cruciate Retaining (CR) Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lagging follow-up.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48
Record Dates: First submitted 2009-08-11; First posted 2009-08-25 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2013-04

CONDITIONS: Arthropathy of Knee
Keywords: Osteoarthritis, traumatic arthritis, avascular necrosis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scorpio® CR Total Knee System (Experimental): Scorpio® CR Total Knee System Study Device
  Interventions: Device: Scorpio® CR Total Knee System

INTERVENTIONS:
Device: Scorpio® CR Total Knee System — All subjects will be implanted with a femoral component, a tibial insert, a tibial tray and a resurfaced patella.
  Other Names: Scorpio® Cruciate Retaining (CR) Total Knee System

SUMMARY:
The purpose of this study is to evaluate the design and functional performance of the Scorpio® Cruciate Retaining (CR) Total Knee System.

DETAILED DESCRIPTION:
The study design is a prospective, multi-center clinical trial. The Scorpio® Cruciate Retaining (CR) Total Knee System is to be implanted for evaluation in this study. This device system is commercially available and is intended for cemented use.

The study group will consist of a maximum of 265 cases, requiring primary total knee replacement, and diagnosed with non-inflammatory arthritis. All subjects will be implanted with a femoral component, a tibial insert, a tibial tray and a resurfaced patella. Subjects receiving bilateral total knee replacements will represent two cases. Study participants will be recruited from 5 institutions.

Subjects will be evaluated preoperatively and at follow-up intervals of 7 wks (± 2 wks), 3 months (± 3 weeks), 6 months (optional visit), 12 months (± 2 months) and annually thereafter (± 2 months). Each subject will be followed for 15 years post-implantation.

The objectives of this study are to:

1. Evaluate the effect of system component design on functional performance.
2. Evaluate the effect of system component design by comparing postoperative functional and radiographic findings with preoperative.
3. Evaluate complications and the rates in which they occur.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or non-pregnant female between the ages of 21-80.
2. The subject requires a primary cemented total knee replacement.
3. The subject has a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
4. The subject has intact collateral ligaments.
5. The subject has signed the IRB approved, study specific Informed Patient Consent Form.
6. The subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient has inflammatory arthritis.
2. The subject is morbidly obese, >60% over ideal body weight for frame and height.
3. The subject has a history of total or unicompartmental reconstruction of the affected joint.
4. Patient has had a high tibial osteotomy or femoral osteotomy.
5. The subject has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
6. The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
7. The subject is immunologically suppressed, or receiving steroids in excess of normal physiological requirements.
8. The subject's bone stock is compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
9. The subject has had a knee fusion to the affected joint.
10. The subject has an active or suspected latent infection in or about the knee joint.
11. The subject is a prisoner.
12. The subject is pregnant.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2001-06; Primary Completion 2009-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Lowry Barnes, MD, Study Chair — Foundation for Musculoskeletal Research and Education; Lawrence Morawa, MD, Principal Investigator — Dearborn Orthopaedics; Arthur Malkani, MD, Principal Investigator — Jewish Physician Group; Frank Kolisek, MD, Principal Investigator — Orthopaedic Research Foundation, Inc.; Steven Harwin, MD, Principal Investigator — Beth Israel Medical Center
Locations (5):
- United States (5):
  - Foundation for Musculoskeletal Research and Education, Little Rock, Arkansas
  - Orthopaedic Research Foundation, Inc., Indianapolis, Indiana
  - Jewish Physician Group, Louisville, Kentucky
  - Dearborn Orthopaedics, Dearborn, Michigan
  - Beth Israel Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 215/229 subjects/cases enrolled and 5 subjects/cases censored=210/224 subjects/cases started
Groups:
- Scorpio® CR Device: All subjects were implanted with the Scorpio® CR Total Knee System Study Device
Period: Overall Study
Arm/Group | Scorpio® CR Device
Started | 210
Completed | 0 (Study was terminated prior to reaching 15 year endpoint.)
Not Completed | 210
Not completed — Death | 7
Not completed — Lost to Follow-up | 22
Not completed — Withdrawal by Subject | 17
Not completed — Unable to return | 1
Not completed — Unwilling to return | 11
Not completed — Intercurrent illness | 1
Not completed — Revision / Removal of Study Implant | 6
Not completed — Overall Study Termination | 145

BASELINE CHARACTERISTICS:
Groups:
- Scorpio® CR Total Knee System Study Device: All subjects were implanted with the Scorpio® CR Knee Arthroplasty Study Device
Arm/Group | Scorpio® CR Total Knee System Study Device
Number analyzed (Participants) | 210
Age, Continuous [Mean (Full Range); unit: years] — For participants who had both knees replaced and enrolled in the study, the age at the time of the first surgery was used.
  One 81 year old participant was enrolled in error and was considered a protocol deviation case, but remained in the study.
  years | 64.46 (8.98) [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 73
Region of Enrollment [Number; unit: participants]
  United States | 210

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Component Design Effect on Functional Knee Society Score and Radiographic Findings.
Description: This study was terminated prior to the protocol defined 15 year endpoint. As such, final outcome measures cannot be posted.
Time Frame: 15 years
Groups:
- Scorpio® CR Device: All subjects received the Scorpio® CR Device
Arm/Group | Scorpio® CR Device
Number analyzed (Participants) | 0

2. Primary Outcome: Evaluate Complication Rate.
Description: as for outcome 1
Time Frame: 15 years
Arm/Group | Scorpio® CR Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: There were a total of 8 serious adverse events reported in 6 subjects.
Arm/Group | Scorpio® CR Total Knee System Study Device
Serious Adverse Events (participants affected / at risk) | 6/210
Other Adverse Events (participants affected / at risk) | 53/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scorpio® CR Total Knee System Study Device (N=210)
Cardiac Disorder (Cardiac disorders) | 1 (1)
Infection and Infestations (Infections and infestations) | 2 (2)
Musculoskeletal and Connective Tissue Disorders (Non-operative site) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and Connective Tissue Disorder (Operative Site) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous System Disorders (Nervous system disorders) | 1 (1)
Vascular Disorders (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scorpio® CR Total Knee System Study Device (N=210)
Musculoskeletal and Connective Tissue Disorders - (Operative Site) (Musculoskeletal and connective tissue disorders) | 53 (68)

LIMITATIONS AND CAVEATS:
This study was terminated early due to lagging follow up prior to the 15 year endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI to publish results of this Clinical Study or the results of the activities hereunder, any abstract, manuscript, presentation or other communication shall be submitted to sponsor for review and approval at least 60 days prior to submission for publication. The sponsor retains the right to deny publication or, at its sole option, to revise the manuscript to delete proprietary or other confidential commercial information.